CLINICAL TRIAL: NCT04256707
Title: Open-Label, Phase 1/2 Study Evaluating the Relative Bioavailability/Bioequivalence of Different Formulations of Selinexor, the Impact of Hepatic Impairment on Selinexor Pharmacokinetics, and the Tolerability and Antitumor Activity of Selinexor Combination Treatment (SPRINT)
Brief Title: Relative Bioavailability/Bioequivalence of Different Formulations of Selinexor, the Impact of Hepatic Impairment on Selinexor Pharmacokinetics, Tolerability and Antitumor Activity of Selinexor Combination Treatment
Acronym: SPRINT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KCP-330-027
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Non-Small Cell Lung Carcinoma (NSCLC); Colorectal Cancer (CRC); Other Solid Tumors
Keywords: Non-small cell lung carcinoma; Selinexor; Docetaxel; Colorectal cancer; KPT-330; Bioequivalence; Relative bioavailability; Pharmacokinetics; Other Solid Tumors
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms | interventions — selinexor; Docetaxel; pembrolizumab; IFL protocol

STUDY DESIGN:
Intervention Model Description: Two part study (monotherapy period and combination therapy period).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Monotherapy: Normal Hepatic Function (Selinexor) (Experimental): (Closed for Enrollment)
  Cohort 1:
  * Week 1: selinexor 5 x 20-mg tablet daily;
  * Week 2: selinexor 1 x 100-mg tablet daily
  Cohort 2:
  * Week 1: selinexor 1 x 100-mg tablet daily;
  * Week 2: selinexor 5 x 20-mg tablet daily.
  Interventions: Drug: Selinexor 100 mg
- Monotherapy: Impaired Hepatic Function (Selinexor) (Experimental): Cohort 3:
  Patients with Moderate Hepatic Impairment with any Solid Tumors;
  - Selinexor 2 x 20-mg tablet once weekly (QW).
  Cohort 4:
  Patients with Severe Hepatic Impairment with any Solid Tumors;
  - Selinexor 2 x 20-mg tablet QW.
  Interventions: Drug: Selinexor 40 mg
- Combination Therapy: NSCLC Arm A: (Selinexor + Docetaxel) (Experimental): (Closed for Enrollment)
  Selinexor 60 mg oral dose QW and docetaxel 75 mg/m^2 intravenously (IV) once every 3 weeks (Non-small cell lung cancer [NSCLC] patients).
  Interventions: Drug: Docetaxel; Drug: Selinexor 60 mg
- Combination Therapy: CRC Arm B: (Selinexor + Pembrolizumab) (Experimental): (Closed for Enrollment)
  Selinexor 80 mg oral does QW and pembrolizumab 200 mg IV every 3 weeks (Colorectal cancer [CRC] Patients).
  Interventions: Drug: Pembrolizumab; Drug: Selinexor 80 mg
- Combination Therapy: CRC Arm C: (Selinexor + FOLFIRI) (Experimental): (Closed for Enrollment)
  Cohort 1:
  Selinexor 40 mg oral dose Days 1, 3, 15 and 18 in a 28-day cycle and FOLFIRI (irinotecan 180 mg/m^2; leucovorin 400 mg/m^2; 5- fluorouracil (5-FU) 400 mg/m^2 bolus then 5-FU 2400 mg/m^2 continuous over 46-48 hours; IV on Day 1 and 15 in a 28-day cycle) (CRC Patients).
  Cohort 2:
  Selinexor 80 mg oral dose Days 1 and 15 in a 28-day cycle and FOLFIRI (irinotecan 180 mg/m^2; leucovorin 400 mg/m^2; 5-FU 400 mg/m^2 bolus then 5-FU 2400 mg/m^2 continuous over 46-48 hours; IV on Day 1 and 15 in a 28-day cycle) (CRC Patients).
  Interventions: Drug: FOLFIRI; Drug: Selinexor 40 mg; Drug: Selinexor 80 mg

INTERVENTIONS:
Drug: Selinexor 100 mg — 100-mg 2 formulations:
  * 5 × 20-mg tablets (Tablet A)
  * 1 × 100-mg tablet (Tablet B)
  Other Names: Xpovio®
  Arms: Monotherapy: Normal Hepatic Function (Selinexor)
Drug: Docetaxel — 75 mg/m^2 IV
  Other Names: Taxotere®
  Arms: Combination Therapy: NSCLC Arm A: (Selinexor + Docetaxel)
Drug: Pembrolizumab — 200 mg IV
  Other Names: Keytruda®
  Arms: Combination Therapy: CRC Arm B: (Selinexor + Pembrolizumab)
Drug: FOLFIRI — FOLFIRI:
  * Irinotecan 180 mg/m^2
  * Leucovorin 400 mg/m^2
  * 5-FU 400 mg/m^2 bolus
  * 5-FU 2400 mg/m^2 IV
  Arms: Combination Therapy: CRC Arm C: (Selinexor + FOLFIRI)
Drug: Selinexor 40 mg — - 2 × 20-mg tablets (Tablet A)
  Other Names: Xpovio®
  Arms: Combination Therapy: CRC Arm C: (Selinexor + FOLFIRI); Monotherapy: Impaired Hepatic Function (Selinexor)
Drug: Selinexor 80 mg — - 4 × 20-mg tablets (Tablet A)
  Other Names: Xpovio®
  Arms: Combination Therapy: CRC Arm B: (Selinexor + Pembrolizumab); Combination Therapy: CRC Arm C: (Selinexor + FOLFIRI)
Drug: Selinexor 60 mg — - 3× 20-mg tablets (Tablet A)
  Other Names: Xpovio®
  Arms: Combination Therapy: NSCLC Arm A: (Selinexor + Docetaxel)

SUMMARY:
This is a Phase 1/2, two-part, multi-arm, open-label study in patients with normal Hepatic Function (HF), with either Non-small cell lung cancer (NSCLC), who have had 1-2 prior lines of treatment, with 1 line containing a checkpoint Inhibitor (CPI); or patients with normal HF, with colorectal cancer (CRC) who have had 1-3 prior lines (KRAS wild-type [WT]) or 1-2 prior lines (mutant KRAS) of treatment with no CPI; or patients with impaired HF, with any solid tumor, who have had at least 1 prior line of treatment.

The study will comprise 2 treatment periods (monotherapy and combination therapy).

The purposes of this study, during Monotherapy period, are: (1) to determine the relative bioavailability of the 100 milligrams (mg) (Tablet B) and 20 mg (Tablet A) tablets of selinexor at 100 mg once weekly (QW) dose in patients with normal hepatic function; and (2) to assess the PK of selinexor after a single dose of 40 mg (2 × 20 mg), among patients with moderate and severe hepatic impairment, relative to 100 mg (5 × 20 mg), among patients with normal hepatic function; and, during the Combination therapy period, to assess the preliminary anti-tumor activity of selinexor in combination with docetaxel in patients with NSCLC and with pembrolizumab or folinic acid, 5-fluorouracil, and irinotecan (FOLFIRI) in patients with CRC.

DETAILED DESCRIPTION:
Up to 120 patients will be enrolled, of which, 20 with normal HF will be able to continue from Monotherapy to Combination therapy and up to 106 patients with normal HF will receive combination therapy in total. Patients with impaired hepatic function can only participate in the Monotherapy part of the study.

Monotherapy Period:

For the Monotherapy Period of Study KCP-330-027, patients with normal hepatic function (n=20), will be allocated to one of two test formulation treatment arms, and will receive a cross-over once weekly oral dosing, with either 1x100 mg or 5x20 mg selinexor, for 2 weeks, and then will have the option to move on to the combination treatment part of the study. Patients with either moderately or severely impaired hepatic functions will be treated with 2x20 mg selinexor weekly (with an option to increase the dose every 3 weeks by 20 mg increments, up to 80 mg).

For the assessment of hepatic impairment, participants with any type of advanced or metastatic solid tumor who have moderate or severe hepatic impairment will be enrolled in Moderate Hepatic Impairment (MHI) (n=8) and Severe Hepatic Impairment (SHI) (n=6) arms, respectively and will be treated with 2 × 20 mg selinexor, weekly.

For Weeks 1 and 2, following an overnight fast of at least 10 hours, patients will be fed a standard low-fat meal 30 minutes prior to administration of once weekly selinexor. Patients should finish the meal in 30 minutes or less; however, selinexor dose should be administered 30 minutes after start of the meal.

Blood sampling for selinexor PK analyses will be collected ≤10 minutes (m) pre selinexor dose, and at 15m (±5m), 30m (±5m), 1 hour (h) (±5m), 1.5h (±5m), 2h (±10m), 3h (±10m), 4h (±10m), 5h (±10m), 6h (±10m), 8h (±20m), 10h (±20m; optional), 24h (±1h), 30h (±1h), and 48h (±2h) post selinexor dose. Practitioners must record the actual clock time for selinexor dose, and each sample drawn.

If a patient experiences emesis during the first 6 hours of the PK sampling, the PK results for that week will be excluded from the PK analysis dataset, and all testing timepoints must be re-collected during the following week (in this case, the same dosing formulation should be repeated on the following week, and other dosing formulation will be given the week after that).

Patients who will complete the Monotherapy Period will be reassessed for continuation to the Combination Therapy Period, as long as their Hepatic Function remains normal.

If a patient experiences significant toxicity related to selinexor and can't start the combination therapy immediately following monotherapy, dose interruption and weekly retesting are allowed for up to 21 days after the end of Monotherapy treatment visit. Patients requiring >21 days to recover from toxicities related to selinexor should be discussed with the Sponsor's Medical Monitor for documented approval to continue to the Combination Therapy Period. Reassessment may be extended then and following Medical Monitor approval up to 28 days.

Combination Therapy Period:

In the combination treatment period of the study, patients with normal hepatic functions will be allocated to one of 3 arms (with Arm C divided into 2 cohorts): Arm A (n= up to 40): Patients with NSCLC who have had up to 2 lines of prior systemic treatment with 1 line containing a CPI will receive 60 mg selinexor weekly, in combination with docetaxel 75 milligrams per meter square (mg/m^2) once every 3 weeks; Arm B (n= up to 40): Patients with CRC (KRAS WT) who have had up to 3 lines of prior systemic treatment or patients with CRC (KRAS mutant [KRAS Mut]) who have had up to 2 lines of prior systemic treatment, with no lines containing a checkpoint inhibitor (CPI) will receive 80 mg selinexor weekly, in combination with pembrolizumab 200 mg once every 3 weeks; Arm C (n<=26): Patients with CRC (regardless of KRAS status) who have had up to 2 lines of prior systemic treatment (regardless of CPI use) will receive either: (Cohort 1) selinexor 40 mg on days 1, 3, 15 and 18 in 28-day cycle + FOLFIRI; or (Cohort 2) selinexor 80 mg on days 1 and 15 in 28-day cycle + FOLFIRI.

Combination Therapy Period Patients will receive combination treatment until progressive disease (PD) or intolerable toxicity.

During both study periods, safety will be assessed through continuous reporting of adverse events (AEs), treatment-emergent adverse events (TEAEs), regularly scheduled clinical laboratory tests (hematologic and chemical), and physical examinations.

Tumor assessment will be performed with either computed tomography (CT) or magnetic resonance imaging (MRI) (CT with contrast preferred; for each patient, the imaging method should remain the same throughout the study).

Following treatment, patients will come in for a safety visit (approximately 30 days after the last dose of combination therapy) and will be followed for up to 2 years after that. Patients who discontinued due to PD will be followed for survival, and patients who discontinued for reasons other than PD will have tumor assessments until PD or until the start of new anti-neoplastic therapy, after which they will be followed for survival.

ELIGIBILITY:
Key Inclusion Criteria:

Common inclusion criteria for all patients:

1. Are greater than or equal to [≥] 18 years of age at the time of informed consent.
2. Have histologically confirmed solid tumor (any type of advanced or metastatic solid tumor for the Hepatic Impairment Arm of the Monotherapy Part), advanced or metastatic NSCLC or CRC and evidence of measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST v1.1).
3. Willing to provide signed written informed consent in accordance with federal, local, and institutional guidelines and comply with all requirements of the study.
4. Female patient of childbearing potential must have a negative serum pregnancy test at screening and agree to use highly effective (dual methods of) contraception throughout the study and for 4 months following the last dose of study drug; and male patients must use an effective barrier method of contraception throughout the study and for 4 months following the last dose of study drug if sexually active. Male patients must agree not to donate sperm during the study treatment period.

   For the Monotherapy Part only (bioavailability/bioequivalence [BA/BE] and hepatic impairment [HI] arms):
5. Have received at least 1 line of systemic anticancer treatment unless there is no first-line standard of care therapy or standard of care therapy is contraindicated adjuvant or neoadjuvant therapy is not counted as one line of systemic therapy). Patients must have failed prior standard curative therapy for their disease, must be intolerant to or be ineligible for any potentially curative approved treatment, irrespective of line of therapy.
6. Must have either normal hepatic function, or moderate or severe hepatic impairment (as defined by the NCI organ dysfunction working group (NCI-ODWG) criteria:

   1. S20-100 and S100-20 arms: normal hepatic function (total bilirubin and aspartate aminotransferase [AST] less than or equal to [≤] upper limit of normal [ULN]).

      Note: Patients with mild hepatic dysfunction (total bilirubin greater than [>] 1 to 1.5 × ULN or AST > ULN) may be included if liver function tests are stable for the past 3 months and enrollment is approved in writing by the Sponsor's Medical Monitor.
   2. MHI arm: ≥1 week of documented moderate hepatic impairment (total bilirubin >1.5-3 × ULN, any level of AST).
   3. SHI arm: ≥1 week of documented severe hepatic impairment (total bilirubin >3-10 × ULN, any level of AST).

   For Combination Therapy Part only:
7. Previous treatment lines (adjuvant or neoadjuvant therapy is not counted as one line of systemic therapy):

   1. Arm A: For patients with NSCLC, have received 1-2 prior lines of systemic anti-cancer treatment with 1 regimen including an anti-PD-1/L1 monoclonal antibody (mAb)
   2. Arm B: For patients with RAS mutant CRC, 1-2 prior lines of systemic treatments, and no prior anti- programmed cell death protein 1/L1 monoclonal antibody (anti-PD-1/L1 mAb).

      * KRAS WT: have 1-3 prior lines of systemic treatments.
      * KRAS mutant (at least 50 percent [%] of patients): 1-2 prior lines of systemic treatments.
   3. Arm C: For patients with CRC participating in the combination arm with FOLFIRI, 1-2 prior lines of systemic therapy are allowed.
   4. Arm B and C in CRC: patient with CRC who are not candidates for curative resection of metastatic lesions.
8. Must have hepatic function as follows:

   1. Arm A (combination with docetaxel): patients with NSCLC who are to receive docetaxel and have bilirubin ≤ ULN, and AST and/or alanine transaminase (ALT) ≤ 1.5 x ULN.
   2. Arm B and C: total bilirubin ≤ 1.5 × ULN and AST ≤ 2.5 x ULN, AST ≤ 2.5 x ULN; for Arm B, unless bilirubin elevation is related to Gilbert's Syndrome for which bilirubin must be ≤ 4 x ULN.

Key Exclusion Criteria:

Common exclusion criteria for all patients:

1. Have inadequate hematopoietic function defined as (without transfusion or growth factor support within 7 days prior to first dose):

   a. absolute neutrophil count (ANC) <1.5 × 109/liter (L); platelet count (PLT) <100 × 109/L; or hemoglobin (Hb) <9 gram per deciliter (g/dL).
2. Have inadequate renal function defined as a calculated creatinine clearance (CrCl) of <20 mL/min using the formula of Cockcroft and Gault.
3. Have any other medical condition especially any gastrointestinal (GI) dysfunctions or GI disease that could interfere with the absorption of selinexor (e.g., inability to swallow or retain oral medications, malabsorption syndrome, a history of GI surgery which may result in intestinal blind loop, significant gastroparesis, unresolved nausea, vomiting, or diarrhea [National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Grade >1]).
4. Ongoing infection requiring parenteral antibiotics, antivirals, or antifungals on Day 1 dosing.
5. Prior exposure to a SINE compound or selinexor.
6. Insufficient time since or not recovered from procedures or anti-cancer therapy, defined as:

   1. Not recovered from major surgery ≤21 days prior to Day 1 dosing. Minor procedures, such as biopsies, dental work, or placement of a port or intravenous (IV) line for infusion are permitted.
   2. Have ongoing clinically significant anti-cancer therapy-related toxicities CTCAE Grade >1. Patients with any of the following will not be excluded: immune checkpoint-related endocrinopathies that are well controlled with hormonal supplements, patients with electrolyte abnormalities that are well-managed with supplementation, patients with Grade 2 lymphopenia, or patients with alopecia of any grade. In specific cases, patients whose toxicity has stabilized or with Grade 2 non-hematologic toxicities can be allowed following documented approval by the Sponsor's Medical Monitor.
   3. Had last dose of previous anti-cancer therapy ≤14 days prior to Day 1 dosing.
   4. Palliative radiotherapy >14 days prior to the study is allowed.
   5. Received investigational drugs in other clinical trials within 28 days, or 5 half-lives of the investigational drug (whichever is shorter), prior to Cycle 1 Day 1 (C1D1).
7. Serious active psychiatric or active medical condition that could interfere with participation in the study or in the opinion of the Investigator would make study involvement unreasonably hazardous.
8. In the opinion of the Investigator, patients who are below their ideal body weight and would be unduly impacted by changes in their weight.
9. Known allergy to selinexor (all patients), docetaxel (NSCLC Arm A only), pembrolizumab (CRC arm B only), OR 5-FU, leucovorin, or irinotecan (CRC Arm C only).
10. Female patients who are pregnant or breastfeeding. For Monotherapy Part only (BA/BE and HI arms):
11. Have an Eastern Cooperative Oncology Group (ECOG) performance status of:

    1. ≥3 for patients to be enrolled into the S20-100 or S100-20 arms of the study.
    2. ≥4 for patients to be enrolled into the MHI and SHI arms of the study.
12. For MHI and SHI arms: ANC <1 × 109/L; PLT <75 × 109/L; or Hb <8 g/dL.
13. Received strong cytochrome P450 3A (CYP3A) inhibitors ≤7 days prior to Day 1 dosing OR strong CYP3A inducers ≤14 days prior to Day 1 dosing.
14. Inability or unwillingness to undergo a series of PK sampling.

    For Combination Therapy Part only:
15. Have an Eastern Cooperative Oncology Group (ECOG) performance status of ≥3 for Arms A and B and ECOG PS ≥2 for Arm C.
16. Arm B patients with CRC who are to receive pembrolizumab:

    1. Had a diagnosis of immunodeficiency or are receiving systemic steroid therapy (>10 milligram per day [mg/day] of prednisone or equivalent) or any other form of immunosuppressive therapy.
    2. Patients with controlled diabetes mellitus and patients with endocrinopathies on stable hormone replacement therapy, are eligible for the trial.
    3. Have active autoimmune disease requiring systemic treatment during the past 2 years. Type 1 diabetes mellitus, hypothyroidism only requiring hormone replacement skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted.

       Note: The Investigator needs to evaluate the patient's medical history to confirm that they are eligible to receive the combination with pembrolizumab per these criteria.
    4. For patients with CRC who have received live-attenuated vaccine against an infectious disease (e.g., nasal spray influenza vaccine) ≤14 days prior to the intended C1D1 of the Combination Therapy.
17. Arm C: Patients with known dihydropyrimidine dehydrogenase (DPD) deficiency. Note: for patients who are initially enrolled onto the BA/BE arm in the monotherapy part and plan to switch to combination therapy after completing the planned dosing and PK sample collection, dose interruption between the Monotherapy Part and the Combination Therapy Part is allowed for recovery from AEs. Patients requiring >21 days to recover from toxicities related to selinexor should be discussed with the Sponsor's Medical Monitor for documented approval to continue to the Combination Therapy Part if inclusion/exclusion criteria are met. Experiencing PD during the Monotherapy Part does not constitute exclusion from the Combination Therapy Part.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Monotherapy Period: Area Under the Concentration-Time Curve from Time Zero to Time of Last Concentration (AUC 0-t) of Selinexor in Patients with Normal, Moderate and Severe Hepatic Function | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 24, 30, and 48 hours post-dose on Days 1 and 8
Monotherapy Period: Area Under the Concentration-Time Curve from Time Zero Extrapolated to Infinity (AUC 0-inf) of Selinexor in Patients with Normal, Moderate and Severe Hepatic Function | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 24, 30, and 48 hours post-dose on Days 1 and 8
Monotherapy Period: Maximum Plasma Concentration (Cmax) of Selinexor in Patients with Normal, Moderate and Severe Hepatic Function | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 24, 30, and 48 hours post-dose on Days 1 and 8
Combination Therapy Period: Arm A and B: Overall Response Rate (ORR) as Assessed by Response Criteria in Solid Tumors Version 1.1 (RECIST 1.1) | Up to 36 months
Combination Therapy Period: Arm C: Number of Patients With Adverse Events (AEs) | From start of study drug administration up to survival follow-up (Up to 36 months)

SECONDARY OUTCOMES:
Monotherapy Period: Time to Maximum Observed Concentration (Tmax) of Selinexor in Patients with Normal, Moderate and Severe Hepatic Impairment | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 24, 30, and 48 hours post-dose on Days 1 and 8
Monotherapy Period: Terminal Elimination Rate Constant (Lambda z) of Selinexor in Patients with Normal, Moderate and Severe Hepatic Impairment | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 24, 30, and 48 hours post-dose on Days 1 and 8
Monotherapy Period: Terminal Half-Life (t1/2) of Selinexor in Patients with Normal, Moderate and Severe Hepatic Impairment | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 24, 30, and 48 hours post-dose on Days 1 and 8
Monotherapy Period: Apparent Clearance (CL/F) of Selinexor in Patients with Normal, Moderate and Severe Hepatic Impairment | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 24, 30, and 48 hours post-dose on Days 1 and 8
Monotherapy Period: Apparent Volume of Distribution (Vd/F) of Selinexor in Patients with Normal, Moderate and Severe Hepatic Impairment | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 24, 30, and 48 hours post-dose on Days 1 and 8
Monotherapy Period: Fraction Unbound (fu) of Selinexor (Tablet A) in Plasma | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 24, 30, and 48 hours post-dose on Days 1 and 8
Monotherapy Period: Maximum Free-Drug Concentration (Cmaxu) of Selinexor (Tablet A) in Plasma | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 24, 30, and 48 hours post-dose on Days 1 and 8
Monotherapy Period: Area Under the Free-Drug Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUCu) of Selinexor (Tablet A) in Plasma | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 24, 30, and 48 hours post-dose on Days 1 and 8
Monotherapy Period: Apparent Free-drug Clearance (CLu/F) of Selinexor (Tablet A) in Plasma | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 24, 30, and 48 hours post-dose on Days 1 and 8
Monotherapy Period: Apparent Free-drug Volume of Distribution (Vu/F) of Selinexor (Tablet A) in Plasma | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 24, 30, and 48 hours post-dose on Days 1 and 8
Combination Therapy Period: Progression-free Survival (PFS): Arms A and C as Assessed by RECIST 1.1 and Arm B as Assessed by iRECIST | Up to 36 months
Combination Therapy Period: Duration of Response (DOR): Arms A and C as Assessed by RECIST 1.1 and Arm B as Assessed by iRECIST | Up to 36 months
Combination Therapy Period: Disease Control Rate (DCR): Arms A and C: as Assessed by RECIST 1.1 and Arm B as Assessed by iRECIST | Up to 36 months
Combination Therapy Period: Overall Survival (OS): Arms A and C as Assessed by RECIST 1.1 and Arm B as Assessed by iRECIST | Up to 36 months
Monotherapy Period: Number of Patients With Adverse Events (AEs) | From start of study drug administration up to survival follow-up (up to 36 months)
Combination Therapy Period: Arm A and B: Number of Patients With Adverse Events (AEs) | From start of study drug administration up to survival follow-up (up to 36 months)
Combination Therapy Period: Arm C: Overall Response Rate (ORR) as Assessed by RECIST 1.1 | Up to 36 months

CONTACTS AND LOCATIONS:
Locations (11):
- Israel (11):
  - Hadassah Ein Karem University Hospital, Jerusalem, Jerusalem
  - University Hospital Assuta Ashdod, Ashdod
  - Soroka University Medical Center, Beersheba
  - Oncology Department Hillel Yaffe Medical Center, Hadera
  - Rambam Health Care Campus, Haifa
  - Shaarei Zedek Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Galilee Medical Center, Nahariya
  - Rabin Medical Center, Petah Tikva
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
  - Sheba Medical Center, Tel Litwinsky

IPD SHARING:
Plan to Share IPD: Undecided